CLINICAL TRIAL: NCT02968355
Title: Clinical Evaluation of the FilmArray® Global Fever (GF) Panel
Status: Completed | Type: Observational
Sponsor: BioFire Defense LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: SDY-017266; HHSN272201600002C (Other Grant/Funding Number: NIAID); W911QY-13-D-0080 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimen may be retained at the participating clinical sites for future use. Specimen nucleic acid may be retained at BioFire and participating clinical sites for future performance evaluations of the FilmArray.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects/Specimens: Subjects/Specimens that meet the eligibility criteria
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study
  Other Names: FilmArray

SUMMARY:
This study will evaluate the clinical sensitivity and specificity of the FilmArray Global Fever (GF) Panel.

DETAILED DESCRIPTION:
The FilmArray Global Fever (GF) Panel, developed by BioFire Defense in collaboration with the U.S. Department of Defense and NIAID, uses an automated, multiplex PCR system to evaluate whole blood samples for 19 pathogens simultaneously in under an hour. Targets of the GF Panel are Chikungunya virus, CCHF virus, dengue virus (serotypes 1-4), Ebolavirus, Lassa virus, Marburgvirus, West Nile virus, Yellow fever virus, Zika virus, Bacillus anthracis, Francisella tularensis, Leptospira spp., Salmonella enterica serovar Typhi and Paratyphi A, Yersinia pestis, Leishmania donovani complex, Plasmodium spp., P. falciparum, and P. ovale/vivax. BioFire Defense is conducting a prospective clinical study to evaluate the sensitivity and specificity of the GF Panel when used to test blood collected from subjects with fever or who have recently had fever. This multi-center study is being conducted at locations around the world.

ELIGIBILITY:
Inclusion Criteria:

* Whole blood in EDTA (prospectively collected via informed consent)
* Subject has a recorded or self-reported fever within the past two days.
* Subject has not participated in the study within the last 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with fever will be prospectively enrolled, and whole blood will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 2084 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of the FilmArray Global Fever (GF) Panel | 18 months
  Percent Positive Agreement and Percent Negative Agreement between FilmArray Result and Comparator Assay

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Phillips, Ph. D., Study Director — BioFire Defense LLC
Locations (11):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - Washington University, St Louis, Missouri
- Naval Medical Research Unit Two, Phnom Penh, Cambodia
- United States Army Medical Research Directorate Georgia, Tbilisi, Georgia
- Naval Medical Research Unit Three, Navrongo, Ghana
- Universidad Nacional Autonoma de Honduras, Tegucigalpa, Central District, Honduras
- United States Army Medical Research Directorate Kenya, Kisumu, Kenya
- Naval Medical Research Unit Six, Iquitos, Peru
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania
- Armed Forces Research Institute of Medical Sciences, Bangkok, Thailand
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Manabe YC, Betz J, Jackson O, Asoala V, Bazan I, Blair PW, Chang A, Chusri S, Crump JA, Edgel KA, Faix DJ, Fernandez S, Fox AT, Garcia JA, Grogl M, Hansen EA, Heang V, House SL, Jongsakul K, Kaburise MB, Klungthong C, Lamorde M, Letizia AG, Lorenzana I, Luy M, Maro VP, Mores CN, Myers CA, Oduro AR, Parham L, Porzucek AJ, Prouty M, Rabiger DS, Rubach MP, Siles C, Silva M, Ukachu C, Waitumbi JN, Phillips CL, Jones BW. Clinical evaluation of the BioFire Global Fever Panel for the identification of malaria, leptospirosis, chikungunya, and dengue from whole blood: a prospective, multicentre, cross-sectional diagnostic accuracy study. Lancet Infect Dis. 2022 Sep;22(9):1356-1364. doi: 10.1016/S1473-3099(22)00290-0. Epub 2022 Jun 15. PMID 35716700

DOCUMENTS (1):
  • Informed Consent Form (2020-03-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02968355/ICF_000.pdf